CLINICAL TRIAL: NCT05515055
Title: Does Relative Hypoglycaemia &/or Sleep Disturbance Contribute to the Lethargy Observed in Addison's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ED22/147142
Record Dates: First submitted 2022-05-19; First posted 2022-08-25 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Addison Disease
MeSH Terms: conditions — Addison Disease | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood test — 1 blood sample extra to standard of care is taken

SUMMARY:
Addison's disease is a condition that leads to a reduction in production of steroid hormones from the adrenal glands. These hormones, particularly cortisol have many important roles in the body, one of which is increasing blood sugar. These steroids will be replaced with tablets but fails to mimic the normal increase in natural cortisol levels which increase from around 2am in the early morning. Furthermore, steroid tablets have been associated with stopping patients from going to sleep.

Patients with Addison's disease on treatment still complain of excessive fatigue and have an increased risk of death from blood vessel diseases. Some case reports have shown some patients with Addison's disease to have low blood sugars overnight.

To investigate the possible causes of fatigue in Addison's disease by examining sugar levels and sleep patterns of our patients. Blood clotting will also be looked at as a potential mechanism for the unexplained increase in blood vessel diseases. To examine sugar levels a small probe will be attached to the upper arm which the patients will wear for 14 days to measure blood glucose very regularly and is painless. Additionally the patients will wear a watch that monitors sleep, movement, and light. A single blood sample will be taken to measure vascular risk markers and how the blood clots.

After wearing the monitors the subjects will complete questionnaires assessing quality of life. Healthy individuals will be recruited to undergo the same monitoring to act as a control group.

The data data obtained between Addison's disease and healthy subjects will be compared.

The scores from the questionnaires will be compared to the glucose and sleep readings to ascertain if there is a link between low blood sugars or sleep disturbance and their quality of life to determine if any physical abnormalities translate in to the poor quality of life.

DETAILED DESCRIPTION:
Patients with primary adrenal insufficiency (PAI) have impaired subjective health status (1, 2) and excess mortality (3, 4). Cardiovascular disease is the greatest contributor towards the excess mortality (3). How current glucocorticoid replacement translates into these adverse sequelea is not understood. Excess and inadequate glucocorticoid replacement likely both contribute. Endogenous cortisol levels rapidly increase from 2am, peaking before waking, and thereafter fall through the day to a nadir around midnight. Hydrocortisone is the preferred glucocorticoid used for replacement therapy in PAI. Current glucocorticoid replacement regimens try to mimic the normal diurnal cortisol rhythm (5). The most commonly used regimens involve use of hydrocortisone (bio-identical to cortisol) administered three times per day (6). As cortisol levels are highest in the morning and fall through the day, a larger dose of hydrocortisone is given on waking with small doses thereafter. It is important in the timing of these doses that there is overlap to avoid periods of cortisol insufficiency. Although regimens aim to replicate the daytime cortisol profile, they cannot currently provide replacement in the early morning hours (2am-7am). This leads to a period of glucocorticoid insufficiency during sleep. Studies using continuous subcutaneous infusion (CSII) of hydrocortisone deliver hydrocortisone in a manner that mimics the normal diurnal rhythm of cortisol, including the period between 2am and waking. Hydrocortisone delivered by CSII has been associated with improvements in well-being in patients with PAI (7), though have not been used in an adequate number of patients for long enough duration to assess the impact on the excess mortality.

Insulin sensitivity is greatest between 2am-4am consequent on the diurnal rhythm of insulin counter-regulatory hormones. Consequently type I diabetic patients are at greatest risk of hypoglycaemia at this time. Glucocorticoid insufficiency increases glucose oxidation and decreases glucose production translating to increased insulin sensitivity. PAI is associated with hypoglycaemic events, though generally in children rather than adults. Using continuous glucose monitoring (CGM) a single case report (8) and a small series identified two patients with nocturnal hypoglycaemia (9). The series did not contain a control group and therefore was unable to determine if nocturnal glucose levels were lower in the patients compared with the normal population.

Furthermore, glucocorticoids have been associated with disruption of sleep, particularly difficulties getting to sleep (10). Therefore taking of replacement hydrocortisone after 6pm in the evening is avoided so that the majority of the hydrocortisone will have been metabolised before the patients retires to sleep. There are however marked differences in the timing of doses of hydrocortisone with patients often taking their doses around other life commitments, or when they are most likely to remember (i.e. first thing in the morning and last thing at night). A significant proportion of patients therefore take their last dose of steroids in the late evening or immediately prior to trying to sleep (6). This can lead hydrocortisone being taken later than prescribed and potentially impacting on sleep. However, as the dose of replacement hydrocortisone is low when given in the evening it is not known if sleep is adversely affected in contrast to that observed with higher therapeutic doses of glucocorticoids?

Finally, much of the excess mortality of patients with primary adrenal insufficiency is reported to relate to vascular disease (3). Vascular risk factors are variably reported to be increased in PAI (11). However, the mechanism by which the excess vascular disease occurs remains incompletely understood.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >18 years
2. Known to have Addison's disease with or without type 1 diabetes
3. They are able to provide valid written consent

Exclusion Criteria:

1. Having significant kidney disease
2. Having active cancer, other than localised/non-aggressive skin cancer
3. Being unable to provide valid written consent
4. Are deemed to be inappropriate to be enrolled in the study by senior members of the research team. This may involve things such as the patient being very frail and struggles to get to and from the hospital, would have problems using the equipment due to significant visual problems or problems with hands or are known to have significant problems with low blood sugars (in those with diabetes) and already take measures to prevent this. Other exclusions may be made at the discretion of the senior investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Importantly healthy people will be recruited who do not suffer from either Addison's disease or diabetes and will undergo the same process as detailed above to act as a healthy control group. The same exclusion criteria will apply to these participants. There are a number of people (termed controls) who have helped the research team with previous studies who will be invited to participate. These controls will be matched to a participant who suffers from Addison's disease/Addison's disease and type 1 diabetes by age, sex and a measure of height and weight termed body mass index (BMI) It is important that the two groups contain a similar population (other than suffering from Addison's disease) so that results are robust and bias is avoided.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of low blood sugars events overnight in patients with Addison's disease will be measured to determine if there is an increased number of low blood sugars events overnight in patients who suffer from Addison's disease. | 3 months

SECONDARY OUTCOMES:
Is the mean blood sugars of patient's with Addison's disease lower than in healthy subjects and Is there greater variation in blood sugar in patients with Addison's disease? | 3 months
Does having low blood sugars contribute to the impaired quality of life of patients with Addison's disease and does sleep disturbance contribute to the impaired quality of life of patients with Addison's disease? | 3 months
To examine vascular risk factors, particularly abnormalities of clot formation and degradation, that may contribute to the reported excess mortality of patients with PAI. | 3 months
Does physiological steroid replacement lead to disturbance of normal sleep patterns? | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No